CLINICAL TRIAL: NCT02645929
Title: Reflective Function as a Mediator of Interpersonal Psychotherapy (IPT) for Posttraumatic Stress Disorder
Brief Title: Reflective Function as a Mediator of Interpersonal Psychotherapy (IPT)
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, John Markowitz, Research Psychiatrist 2; Professor of Clinical Psychiatry, New York State Psychiatric Institute
Other Study IDs: 7211
Record Dates: First submitted 2016-01-03; First posted 2016-01-05 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy (IPT) — IPT is a 14 week psychotherapy for PTSD. SSRF is a brief interview to assess emotional understanding of one's symptoms.

SUMMARY:
Our recent randomized controlled trial of psychotherapies for posttraumatic stress disorder (PTSD) showed that Interpersonal Psychotherapy (IPT) benefitted patients. The mechanism of action for IPT is unclear; unlike most PTSD therapies, it does not work through exposure to trauma reminders. This assessment study will assess Symptom-Specific Reflective Function, a measure of emotional awareness of one's PTSD symptoms, as a potential mediator of IPT, capitalizing on naturalistic treatment of military veterans with PTSD at Columbia University/New York State Psychiatric Institute.

DETAILED DESCRIPTION:
In a randomized controlled study, the investigators recently showed that fourteen weeks of treatment with Interpersonal Psychotherapy (IPT) worked at least as well as the best studied exposure therapy in relieving symptoms of posttraumatic stress disorder (PTSD) (American Journal of Psychiatry, 2015). The investigators do not know the mechanism by which IPT works, however, except that it does not work through exposing patients to reminders of their trauma, as most exposure therapies for PTSD do. Rather, IPT seems to work in part by helping numbed patients to reconnect with and to understand their feelings, then use those feelings to handle interpersonal encounters with other people. One promising measure of this possible mechanism of IPT is Reflective Function, which has two components.

Reflective Functioning (RF) measures how well an individual understands his or her emotions as well as the emotions of significant other people in his or her life. A separate aspect is Symptom-Specific Reflective Function (SSRF), which gauges the individual's emotional understanding of his or her PTSD symptoms. Both RF and SSRF can be measured in a tape recorded interview that takes about 20 minutes, in which the interviewer asks the patient to describe relationships with important people in the patient's life, as well as questions about the patient's understanding of his or her symptoms. The tape is then transcribed for scoring.

A Veterans Clinic at New York State Psychiatric Institute to treat armed service veterans and their families who have PTSD and other psychiatric disorders has opened. This clinic is covered under a separate IRB protocol. As some of the patients in that clinic will receive treatment with IPT, the investigators propose to assess RF, SSRF, and a related measure, the Structured Clinical Interview for Separation Anxiety Symptoms (SCI-SAS), at three points in treatment (before treatment starts; at week 4; and after treatment ends, at week 14) to see whether change in SSRF in particular accounts for improvement in PTSD as measured by the Clinician-Administered PTSD Scale (CAPS), which will be assessed pre-treatment (week 0), mid-treatment (week 7), and post-treatment (week 14). Both veterans and their family members will be eligible for this protocol so long as they meet study eligibility criteria. Because there is no reason to expect that psychotropic medication alters RF, patients who are taking stable doses of medication will be allowed to continue them during IPT treatment.

ELIGIBILITY:
Inclusion Criteria: Method of Ascertainment:

1. Age 18 and older History
2. Primary diagnosis of DSM-5 PTSD Clinical interview: CAPS-5
3. Significant distress affecting social/ occupational functioning Clinical interview, self-report measures PHQ-9, GAD-7, PCL-5, DRRI-2
4. Prior military service (for veteran) or significant relationship with individual with prior military service (for family member) History
5. Able to give consent, fluent in English or Spanish Clinical assessment

Exclusion Criteria:

1. History of Axis I psychiatric diagnosis of psychotic disorder, bipolar disorder, antisocial personality disorder Clinical assessment
2. Unstable or life threatening medical condition Clinical assessment
3. Acute suicide or homicide risk Clinical assessment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 US veterans or their family members suffering from DSM-5 PTSD
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-04; Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | 14 weeks
  The CAPS-5 is the standard measure for PTSD symptom severity

SECONDARY OUTCOMES:
Structured Clinical Interview for Separation Anxiety Symptoms (SCI-SAS) | Administered at study weeks 0, 4, and 14
  This measure of separation anxiety is a proxy for attachment dysregulation.

CONTACTS AND LOCATIONS:
Overall Officials: John C Markowitz, M.D., Principal Investigator — New York State Psychiatric Institute/Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No. We will be happy to release anonymized group data, beginning with its publication.

REFERENCES:
- [Background] Markowitz JC, Petkova E, Neria Y, Van Meter PE, Zhao Y, Hembree E, Lovell K, Biyanova T, Marshall RD. Is Exposure Necessary? A Randomized Clinical Trial of Interpersonal Psychotherapy for PTSD. Am J Psychiatry. 2015 May;172(5):430-40. doi: 10.1176/appi.ajp.2014.14070908. Epub 2015 Feb 13. PMID 25677355
- [Background] Rudden MG, Milrod B, Meehan KB, Falkenstrom F. Symptom-specific reflective functioning: incorporating psychoanalytic measures into clinical trials. J Am Psychoanal Assoc. 2009 Dec;57(6):1473-8. doi: 10.1177/00030651090570060804. No abstract available. PMID 20068250
- [Background] Bovin MJ, Marx BP, Weathers FW, Gallagher MW, Rodriguez P, Schnurr PP, Keane TM. Psychometric properties of the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (PCL-5) in veterans. Psychol Assess. 2016 Nov;28(11):1379-1391. doi: 10.1037/pas0000254. Epub 2015 Dec 14. PMID 26653052
- [Result] Markowitz JC, Milrod B, Luyten P, Holmqvist R. Mentalizing in Interpersonal Psychotherapy. Am J Psychother. 2019 Dec 1;72(4):95-100. doi: 10.1176/appi.psychotherapy.20190021. Epub 2019 Nov 22. PMID 31752509
- [Result] Markowitz JC, Lowell A, Milrod BL, Lopez-Yianilos A, Neria Y. Symptom-Specific Reflective Function as a Potential Mechanism of Interpersonal Psychotherapy Outcome: A Case Report. Am J Psychother. 2020 Mar 1;73(1):35-40. doi: 10.1176/appi.psychotherapy.20190026. Epub 2020 Jan 6. No abstract available. PMID 31902227
- [Result] Milrod B, Keefe JR, Choo TH, Arnon S, Such S, Lowell A, Neria Y, Markowitz JC. Separation anxiety in PTSD: A pilot study of mechanisms in patients undergoing IPT. Depress Anxiety. 2020 Apr;37(4):386-395. doi: 10.1002/da.23003. Epub 2020 Feb 25. PMID 32097526
- See also: Columbia PTSD and trauma website — http://columbiapsychiatry.org/researchclinics/center-trauma-resilience